CLINICAL TRIAL: NCT03709303
Title: Motivations, Expectations, and Decision-making of Sickle Cell Patients in Clinical Research
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 190004; 19-CC-0004
Record Dates: First submitted 2018-10-16; First posted 2018-10-17 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Sickle Cell Disease
Keywords: Informed Consent; Stem Cell Transplantation; Understanding; Optimism; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- SCD patients: Patients with sickle cell disease who have decided about enrollment in an NIH study of PBSCT or Gene therapy

SUMMARY:
Background:

Sickle cell disease is an inherited blood disorder. People with this disease have a problem with their hemoglobin. That is a protein in red blood cells that carries oxygen in the body. Some people with this disease are enrolled in research at NIH. Researchers want to learn more about the thoughts and opinions of those people. This may improve the way researchers explain clinical studies, risks, and benefits to people with the disease.

Objective:

To learn about the motivations, decisions, and experiences in clinical research of people with sickle cell disease.

Eligibility:

Adults ages 18 and older who have sickle cell disease. They must be in an NIH study on this condition. They must have been invited to join either a gene therapy or peripheral blood stem cell transplantation study.

Design:

Participants will have 1 interview. It will be done in a quiet room in the NIH Clinical Center or by video call. It will take about 60 minutes.

The interview will be audio-recorded if the participant agrees.

Participants will be asked about:

* Their experiences with and thoughts on sickle cell disease
* Their decision to participate in clinical research
* Factors that may have affected their decision to participate. These may include family, disease history, or faith.

Participants may complete a few brief questionnaires.

DETAILED DESCRIPTION:
Clinical trials testing potentially curative interventions for sickle cell disease - such as gene therapy (GT) or peripheral blood stem cell transplantation (PBSCT) - have created a novel opportunity for patients with sickle cell disease, for whom standard therapies can only manage but not cure their conditions. But some of these experimental interventions may pose risk of significant adverse events. As the development of these interventions create a new decision-making situation for persons with longstanding diseases, these trials raise questions about the expectations and decision- making process of patients considering and/or participating in them. Given the longstanding debate in the bioethics literature about whether patients expressions of desire for benefit are (1) evidence of false hopes or poor understanding of risks and benefits, or, instead (2) expressions of natural optimism compatible with valid informed consent, these patients present an opportunity to learn about how they make their participation decisions which in turn could inform this longstanding debate.

This study aims to explore the expectations, understanding, motivations, and decision-making of patients with sickle cell disease who have either chosen or declined to enroll in research studies testing experimental interventions. The aim is to better understand how these patients understand the research study, assess risks and benefits at the time of enrollment, make decisions, and react to their health outcomes. As faith and religion are known to play an important part in the lives of persons with sickle cell disease, we will also explore the role of religion and faith in sickle cell patients decision-making and retrospective perspective on their decision.

Primary Hypothesis:

This is a descriptive, explorative study. It may generate hypotheses for future studies.

Purpose of the Study Protocol:

To describe how patients with sickle cell disease understand and make decisions about participating in gene therapy (GT) or peripheral blood stem cell transplantation (PBSCT) clinical trials to shed light about the ethically salient issues regarding enrollment and participation in high- risk, high-reward clinical trials. This information may inform practices around the informed consent process and help researchers better understand the role of family and religion/faith in clinical research decision making.

ELIGIBILITY:
* INCLUSION CRITERIA:

Our inclusion criteria for study subjects are:

* Adult (18+ years and older)
* Sickle cell disease patients who are enrolled in at least one of the following sickle cell disease protocols at the National Institutes of Health, National Heart, Lung, and Blood Disease:

  * Screening study: 08-H-0156
  * Natural history protocol: 04-H-0161
  * PBSCT: 09-H-0225, 17-H-0069, 14-H-0077, 03-H-0170
  * GT: 14-H-0155
* Have made a decision regarding participation in one of the GT or PBSCT protocols (e.g. someone could still be enrolled in Screening study, have made a decision, but not yet enrolled in or have declined enrollment in the GT or PBSCT studies)
* Study subjects will be recruited in two groups: 1) pre-transplant or pre-initiation of gene therapy, including both those who decide to enroll and those who declined to enroll; and 2) post-transplantation or post-GT, including those who had an unsuccessful and those who had a successful transplantation or response to GT.

EXCLUSION CRITERIA:

Study subjects will be excluded if they:

* Lack cognitive capacity
* Are not English speaking
* Have not made a decision about participation in one of the GT or PBSCT protocols for which they are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample will be selected from among SCD patients enrolled in NHLBI protocols at NIH
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Expectations, understanding and motivations for enrollment | Before or after enrollment in PBSCT or GT trial, but after decision made
  Understanding, expectations, motivations, and decision making process

SECONDARY OUTCOMES:
Explore the role of family and religion | After decision made about enrollment
  Description of the role of family, culture, and religion in enrollment decision making

CONTACTS AND LOCATIONS:
Overall Officials: Christine Grady, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kim SY, De Vries R, Holloway RG, Kieburtz K. Understanding the 'therapeutic misconception' from the research participant's perspective. J Med Ethics. 2016 Aug;42(8):522-3. doi: 10.1136/medethics-2016-103597. Epub 2016 May 4. No abstract available. PMID 27145809
- [Background] Pentz RD, White M, Harvey RD, Farmer ZL, Liu Y, Lewis C, Dashevskaya O, Owonikoko T, Khuri FR. Therapeutic misconception, misestimation, and optimism in participants enrolled in phase 1 trials. Cancer. 2012 Sep 15;118(18):4571-8. doi: 10.1002/cncr.27397. Epub 2012 Jan 31. PMID 22294385
- [Background] Adegbola M. Spirituality, Self-Efficacy, and Quality of Life among Adults with Sickle Cell Disease. South Online J Nurs Res. 2011 Apr;11(1):5. PMID 21769284
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-CC-0004.html